CLINICAL TRIAL: NCT00503217
Title: Effect of GnRH Agonist Administration at the Time of Implantation in Intrauterine Insemination Cycles: A Randomized Controlled Trial
Brief Title: GnRH Agonist and Intrauterine Insemination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Bellver, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: VLC-JB-0205-307-9
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Intrauterine Insemination
Keywords: intrauterine insemination; GnRH agonist; implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tryptorelin

SUMMARY:
The aim of this study is to assess whether GnRH agonist administration in the luteal phase improves pregnancy outcome in intrauterine insemination (IUI) cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women < 38 years old
* Bilateral tubal patency confirmed by hysterosonography
* Normal ultrasound scan of uterus and ovaries
* Normal day 3 basal hormones
* Motile sperm count after capacitation ≥ 3 mill/ml

Exclusion Criteria:

* Endometriosis
* Polycystic ovary syndrome
* Uterine disease (polyps, myomas and müllerian diseases)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bellver, MD, Principal Investigator — Instituto Valenciano de la Infertilidad; Elena Labarta, MD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Valencia, Spain